CLINICAL TRIAL: NCT00325299
Title: Magnesium After Alcohol Withdrawal Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finnish Foundation for Alcohol Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFAS-02
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2006-05-12 (Estimated); Status verified 2006-05

CONDITIONS: Alcohol-Induced Disorders
MeSH Terms: conditions — Alcohol-Induced Disorders | interventions — Magnesium

INTERVENTIONS:
Drug: Magnesium

SUMMARY:
The primary purpose is to see if magnesium tablet supplementation will decrease elevated GGT enzyme activity in alcoholic patients immediately after they had been treated for alcohol withdrawal. The secondary aims are to find out whether supplementation decreases the activity of ASAT and ALAT enzymes, increases muscle strength, decreases blood pressure and decreases depressive symptoms among these patients.

DETAILED DESCRIPTION:
Magnesium (Mg) deficiency is common among alcoholics. Animal studies have shown that magnesium deficiency aggravates the hepatic damage caused by alcohol. One study on chronic alcoholics suggested that magnesium supplementation over six weeks decreases abnormally high activities of three enzymes related to liver function: serum gamma-glutamyltransferase (GGT), aspartate-aminotransferase (ASAT) and alanine-aminotransferase (ALAT), and increases muscle strength [4]. These results were, however, significant at the 5% level only when a 1-sided test was applied. It seems that magnesium supplementation may improve liver recovery after a drinking bout, but the evidence is not yet strong enough to warrant clear recommendations for clinical practice. Magnesium deficiency may also be one of the symptoms of depression and may aggravate hypertension. The primary purpose of the present randomized, parallel group, double blind trial is to see if oral magnesium supplementation will decrease elevated GGT enzyme activity in alcoholic patients immediately after they had been treated for alcohol withdrawal. The secondary aims are to find out whether supplementation decreases the activity of ASAT and ALAT enzymes, increases muscle strength, decreases blood pressure and decreases depressive symptoms among these patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to treatment because of an acute alcohol withdrawal
* Elevated serum GGT (men>80, women >50)
* Age 20-64 years
* Fixed address and a telephone to facilitate follow-up

Exclusion Criteria:

* Mg supplementation within the past two months ten 250 mg tablets or more
* History of heart rhythm disturbances
* Contraindications against Mg treatment
* Abnormally high serum creatinine

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178
Dates: Study Completion 2005-09

PRIMARY OUTCOMES:
Serum gamma-glutamyltransferase (GGT) activity

SECONDARY OUTCOMES:
Aspartate-aminotransferase (ASAT) activity
Alanine-aminotransferase (ALAT) activity
Depressive symptoms
Blood pressure
Handgrip muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Kari Poikolainen, Dr Med Sci, Principal Investigator — Finnish Foundation for Alcohol Studies
Locations (1):
- Finnish Foundation for Alcohol Studies, Helsinki, Finland

REFERENCES:
- [Derived] Poikolainen K, Alho H. Magnesium treatment in alcoholics: a randomized clinical trial. Subst Abuse Treat Prev Policy. 2008 Jan 25;3:1. doi: 10.1186/1747-597X-3-1. PMID 18218147